CLINICAL TRIAL: NCT02115373
Title: A Multicenter, Single Arm, Phase Ib/II Study to Evaluate Efficacy, Safety, and PK of MSC2156119J as Monotherapy in Subjects With MET+ Advanced Hepatocellular Carcinoma With Child Pugh Class A Liver Function Who Have Failed Sorafenib Treatment
Brief Title: c-Met Second-Line Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200095_005; 2013-002053-30 (EudraCT Number)
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Results first posted 2019-08-09 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; c-Met inhibitor; Phase 1b; Sorafenib; MSC2156119J
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tepotinib

ARMS (3):
- Phase 1b: Tepotinib 300 mg (Experimental)
  Interventions: Drug: Tepotinib
- Phase 1b: Tepotinib 500 mg (Experimental)
  Interventions: Drug: Tepotinib
- Phase 2: Tepotinib 500 mg (Experimental)
  Interventions: Drug: Tepotinib

INTERVENTIONS:
Drug: Tepotinib — Participants received a single oral dose of Tepotinib 300 milligram (mg) in each 21 days treatment cycle until progressive disease, intolerable toxicity, death, or withdrawal from treatment.
  Other Names: MSC2156119J
  Arms: Phase 1b: Tepotinib 300 mg
Drug: Tepotinib — Participants received a single oral dose of Tepotinib 500 mg daily in each 21 days treatment cycle until progressive disease, intolerable toxicity, death, or withdrawal from treatment.
  Other Names: MSC2156119J
  Arms: Phase 1b: Tepotinib 500 mg; Phase 2: Tepotinib 500 mg

SUMMARY:
This is a Phase 1b/2, multicenter, single arm trial to assess the efficacy, safety, and pharmacokinetics (PK) of MSC2156119J as monotherapy in subjects with MET+ advanced hepatocellular carcinoma (HCC) with child Pugh Class A liver function who have failed sorafenib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HCC
* Child Pugh Class A liver function score
* For Phase 2 only: MET+ status
* Male or female, 18 years of age or older
* Measurable disease in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 (inclusive)
* Availability of a pretreatment tumor biopsy (excluding fine needle aspiration and cytology samples) taken after the subject has discontinued sorafenib and within 28 days before the day of first dosing with MSC2156119J. From the pretreatment biopsy either a formalin-fixed (formalin fixation is mandatory) paraffin-embedded block with tumor tissue (preferred) or at least 15 unstained slides must be sent to the central laboratory prior to enrollment. An associated pathology report must also be sent with the sample
* Previously treated with sorafenib for greater than or equal to 4 weeks and discontinued sorafenib treatment at least 14 days prior to Day 1 due to either intolerance or radiographic progression
* Signed and dated informed consent indicating that the subject (or legally acceptable representative if applicable by local laws) has been informed of all the pertinent aspects of the trial prior to enrollment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other trial procedures
* Life expectancy of at least 3 months as judged by the investigator

Exclusion Criteria:

* Prior systemic anticancer treatment for advanced HCC (except for sorafenib as described in the inclusion criteria)
* Prior treatment with any agent targeting the hepatocyte growth factor (HGF)/c-Met pathway
* Local-regional therapy within 4 weeks before Day 1
* Impaired cardiac function
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-05-18 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center located in, Darmstadt, Germany

REFERENCES:
- [Derived] Xiong W, Hietala SF, Nyberg J, Papasouliotis O, Johne A, Berghoff K, Goteti K, Dong J, Girard P, Venkatakrishnan K, Strotmann R. Exposure-response analyses for the MET inhibitor tepotinib including patients in the pivotal VISION trial: support for dosage recommendations. Cancer Chemother Pharmacol. 2022 Jul;90(1):53-69. doi: 10.1007/s00280-022-04441-3. Epub 2022 Jun 30. PMID 35771259
- [Derived] Decaens T, Barone C, Assenat E, Wermke M, Fasolo A, Merle P, Blanc JF, Grando V, Iacobellis A, Villa E, Trojan J, Straub J, Bruns R, Berghoff K, Scheele J, Raymond E, Faivre S. Phase 1b/2 trial of tepotinib in sorafenib pretreated advanced hepatocellular carcinoma with MET overexpression. Br J Cancer. 2021 Jul;125(2):190-199. doi: 10.1038/s41416-021-01334-9. Epub 2021 Apr 6. PMID 33824476
- See also: : Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant signed informed consent:18 May 2014, Last participant last visit: 14th Feb 2018
Pre-assignment Details: In Phase 1b, 24 participants were screened of which, 17 started the treatment. In Phase 2 ,155 participants were screened, of which 49 participants started the treatment.
Groups:
- Phase 1b: Tepotinib 300 mg: Participants received a single oral dose of Tepotinib 300 milligram (mg) daily in each 21 days treatment cycle until progressive disease, intolerable toxicity, death, or withdrawal from treatment.
- Phase 1b: Tepotinib 500 mg; Phase 2: Tepotinib 500 mg: Participants received a single oral dose of Tepotinib 500 mg daily in each 21 days treatment cycle until progressive disease, intolerable toxicity, death, or withdrawal from treatment.
Period: Overall Study
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
Started | 4 | 13 | 49
Completed | 4 | 13 | 49
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J).
Groups:
- Phase 1b: Tepotinib 300 mg: Participants received a single oral dose of Tepotinib 300mg daily in each 21 days treatment cycle until progressive disease, intolerable toxicity, death, or withdrawal from treatment.
- Phase 1b: Tepotinib 500 mg: Participants received a single oral dose of Tepotinib 500mg daily in each 21 days treatment cycle until progressive disease, intolerable toxicity, death, or withdrawal from treatment.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg | Total
Number analyzed (Participants) | 4 | 13 | 49 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 21 | 25
  >=65 years | 3 | 10 | 28 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 8 | 12
  Male | 2 | 11 | 41 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 1 | 8 | 26 | 35
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 3 | 4 | 20 | 27

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants Experiencing Dose Limiting Toxicity (DLT) According to National Cancer Institute Common Toxicity Criteria (NCI-CTCAE) for Adverse Events (AEs) Version 4.0
Description: DLT: defined using NCI-CTCAE for AEs Version 4.0, as any of following toxicities: Grade 4 neutropenia for more than 7 days; greater than or equal to (>=) Grade 3 febrile neutropenia for more than 1 day; Grade 4 or Grade 3 thrombocytopenia with nontraumatic bleeding; >=Grade 3 uncontrolled nausea/vomiting and/or diarrhoea despite adequate treatment for more than 3 days; >=Grade 3 any non-hematological AE. (DLT defined specifically for following cases: >=Grade 3 liver AE requiring recovery period of more than 7 days or to Grade 1 or less or Grade 2 with liver metastases ; >=Grade 3 lipase and/or amylase elevation with confirmation of pancreatitis. An isolated lipase and/or amylase elevation of >=Grade 3 without clinical/radiological evidence of pancreatitis was not classified as DLT); and AEs assessed by investigators to be exclusively related to the participant's underlying disease or medical condition/concomitant treatment are not considered as DLTs.
Time Frame: Day 1 to Day 21 of Cycle 1 (each cycle was 21 days)
Population: DLT analysis set included all participants who completed Cycle 1 and who received 80 percent (%) or more of the planned cumulative dose of Tepotinib (MSC2156119J) in Cycle 1, and participants who experienced a DLT during Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 11
Participants | 0 | 0

2. Primary Outcome: Phase 2: Number of Participants Who Were Progression-free at 12 Weeks (PFS Status) as Assessed by the Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS status was evaluated by the number of participants who were progression-free at 12 weeks according to RECIST Version 1.1. Participants were considered to be progression-free if the participant had a tumor assessment of Complete Response (CR) defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 millimeter (mm). Partial response (PR) defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters, or Stable Disease (SD) defined as any cases that do not qualify for either partial response or progressive disease (an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started)12 weeks after start of treatment or later.
Time Frame: At 12 weeks post first-dose in Phase 2
Population: Intent to Treat (ITT) set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J). The outcome measure was planned to be analyzed for Phase 2 only.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2: Tepotinib 500 mg: Participants received a single oral dose of Tepotinib 500 mg daily in each 21 day treatment cycle until confirmed disease progression.
Arm/Group | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 49
Participants | 31

3. Secondary Outcome: Phase 1b and Phase 2: Time to Progression According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: TTP was the time (in months) from the date of first study drug administration to the date of radiological confirmation of PD performed according to RECIST Version 1.1. PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started. The descriptive data represents the number of participants with progression.
Time Frame: Time from first study drug administration to the date of first occurrence of radiological progressive disease (PD), assessed up to 12 months after last participant's first dose (assessed maximum up to 1369 days)
Population: ITT set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J).
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Tepotinib 300 mg: Participants received a single oral dose of Tepotinib 300 mg daily in each 21 days treatment cycle until progressive disease, intolerable toxicity, death, or withdrawal from treatment.
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 4 | 13 | 49
Participants | 3 | 9 | 36
Statistical Analysis 1: Comparison: Phase 1b: Tepotinib 300 mg vs Phase 1b: Tepotinib 500 mg; Test type: Other; Median = 2.07, 90% CI 2-sided [1.446 to 7.195] — TTP in months was calculated for Phase 1b: Tepotinib 300 mg and Phase 1b: Tepotinib 500 mg combined
Statistical Analysis 2: Comparison: Phase 2: Tepotinib 500 mg; Test type: Other; Median = 3.98, 90% CI 2-sided [2.858 to 4.238] — TTP in months was calculated for Phase 2: Tepotinib 500 mg

4. Secondary Outcome: Phase 1b and Phase 2: Progression-free Survival (PFS) Time According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS time was defined as the time from date of randomization until date of the first observation of progressive disease (PD) or death due to any cause within 12 weeks of the last tumor assessment in the absence of documented PD, whichever occurs first. PFS was assessed as per RECIST v1.1 as adjudicated by independent endpoint review committee (IERC). PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started. The descriptive data represents number of participants with death or progressive disease.
Time Frame: From randomization up to first observation of PD or death, assessed maximum up to 1369 days
Population: ITT analysis set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 4 | 13 | 49
Participants | 4 | 12 | 38
Statistical Analysis 1: Comparison: Phase 1b: Tepotinib 300 mg vs Phase 1b: Tepotinib 500 mg; Test type: Other; Median = 1.51, 90% CI 2-sided [1.413 to 3.680] — PFS time in months was calculated for Phase 1b: Tepotinib 300 mg and Phase 1b: Tepotinib 500 mg combined
Statistical Analysis 2: Comparison: Phase 2: Tepotinib 500 mg; Test type: Other; Median = 3.22, 90% CI 2-sided [0.03 to 16.53] — PFS time in months was calculated for Phase 2: Tepotinib 500 mg

5. Secondary Outcome: Phase 1b and Phase 2: Progression-free Survival (PFS) Time According to Modified Response Evaluation Criteria in Solid Tumors (mRECIST) for Hepatocellular Carcinoma (HCC)
Description: PFS time was defined as the time from date of randomization until date of the first observation of progressive disease (PD) or death due to any cause within 12 weeks of the last tumor assessment in the absence of documented PD, whichever occurs first. PFS was assessed as per mRECIST for HCC as adjudicated by independent endpoint review committee (IERC). PD was defined as an increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started. The descriptive data represents number of participants with death or progressive disease.
Time Frame: From randomization up to first observation of PD or death, assessed maximum up to 1369 days
Population: ITT analysis set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 4 | 13 | 49
Participants | 4 | 9 | 37
Statistical Analysis 1: Comparison: Phase 1b: Tepotinib 300 mg vs Phase 1b: Tepotinib 500 mg; Test type: Other; Median = 1.48, 90% CI 2-sided [1.413 to 3.844] — PFS time in months was calculated for Phase 1b: Tepotinib 300 mg and Phase 1b: Tepotinib 500 mg combined
Statistical Analysis 2: Comparison: Phase 2: Tepotinib 500 mg; Test type: Other; Median = 3.35, 90% CI 2-sided [2.760 to 4.172] — PFS time in months was was calculated for Phase 2: Tepotinib 500 mg

6. Secondary Outcome: Phase 2: Time-to-symptomatic Progression (TTSP)
Description: Time-to-symptomatic progression was defined as time (in months) from first study drug administration to the date of deterioration of symptoms assessed by Functional Assessment of Cancer Therapy Hepatobiliary Symptom Index 8 (FHSI-8) (defined as at least a 4-point increase, i.e., higher score, compared with baseline value), or deterioration to Eastern Cooperative Oncology Group (ECOG) performance score 4, or death. FHSI-8 assesses hepatobiliary cancer symptoms with total score ranges from 0 to 32 (0 = the best quality of life; 32 = the worst quality of life with severe symptoms). ECOG assess participant's performance status on a scale of 0 to 5, where 0=fully active and 5=dead.
Time Frame: From date of randomization up to 1369 days
Population: ITT analysis set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J). Here, Overall number of participants analyzed signified those participants who had symptomatic progression. As per planned analysis, data for this outcome was analyzed for Phase 2 only.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 41
months | 4.86 [0.03 to 17.97]

7. Secondary Outcome: Phase 1b and Phase 2: Overall Survival (OS) Time
Description: The OS time was defined as the time from randomization to the date of death. The participants who were still alive at the time of data analysis or who were lost to follow-up OS time was censored at the last recorded date that the participant was known to be alive before the data cutoff date. The descriptive data represents number of participants who had an event of death.
Time Frame: From date of randomization up to the date of death, assessed maximum up to 1369 days
Population: ITT analysis set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 4 | 13 | 49
Participants | 3 | 11 | 40
Statistical Analysis 1: Comparison: Phase 1b: Tepotinib 300 mg vs Phase 1b: Tepotinib 500 mg; Test type: Other; Median = 7.20, 90% CI 2-sided [3.680 to 10.119] — Overall Survival time in months was calculated for Phase 1b: Tepotinib 300 mg and Phase 1b: Tepotinib 500 mg combined
Statistical Analysis 2: Comparison: Phase 2: Tepotinib 500 mg; Test type: Other; Median = 5.55, 90% CI 2-sided [5.092 to 8.181] — Overall Survival time in months was calculated for Phase 2: Tepotinib 500 mg

8. Secondary Outcome: Phase 1b and Phase 2: Percentage of Participants With Best Overall Tumor Assessment of CR or PR According to RECIST v1.1
Description: Percentage of participants with best overall tumor assessment of (CR or PR) according to RECIST Version 1.1 was reported. CR defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started.
Time Frame: From date of randomization up to first occurrence of PD, assessed maximum up to 1369 days
Population: ITT analysis set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J).
Measure: Number (90% Confidence Interval); unit: percentage of Participants
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 4 | 13 | 49
percentage of Participants | 50.0 [9.8 to 90.2] | 0.0 [0.0 to 20.6] | 8.2 [2.8 to 17.7]

9. Secondary Outcome: Phase 1b and Phase 2: Percentage of Participants With Disease Control
Description: Disease control was defined as CR, PR, or SD as the best overall response according to RECIST Version 1.1. Complete Response (CR) defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial response (PR) defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters, or Stable Disease (SD) defined as any cases that do not qualify for either partial response or progressive disease (an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started)12 weeks after start of treatment or later. Percentage of Participants With Disease Control were reported.
Time Frame: From date of randomization up to first occurrence of PD, assessed maximum up to 1369 days
Population: ITT analysis set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J).
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 4 | 13 | 49
percentage of participants | 50.0 [9.8 to 90.2] | 30.8 [11.3 to 57.3] | 57.1 [44.4 to 69.2]

10. Secondary Outcome: Phase 1b and Phase 2: Percentage of Participants With Biological Response
Description: Percentage of participants with biological response was measured by serum Alpha-Fetoprotein (AFP), defined as a greater than 20% decrease in AFP level by Cycle 3 (each cycle is of 21 days) compared with baseline.
Time Frame: Baseline up to Cycle 3 (each cycle is 21 days)
Population: ITT analysis set included all participants who had been administered at least one dose of Tepotinib (MSC2156119J). Here, "Overall number of participants analyzed" signified the participants with baseline and post baseline AFP assessments.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1b: Tepotinib 300 mg: Participants received a single oral dose of Tepotinib 300 mg daily in each 21 day treatment cycle until confirmed disease progression.
- Phase 1b: Tepotinib 500 mg; Phase 2: Tepotinib 500 mg: Participants received a single oral dose of Tepotinib 500 mg daily in each 21 day treatment cycle until confirmed disease progression.
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 11 | 45
percentage of participants | 66.7 [13.5 to 98.3] | 45.5 [20.0 to 72.9] | 31.1 [19.9 to 44.3]

11. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Tepotinib
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours Post-dose on Day 1 and Day 15 of Treatment Cycle 1 (each cycle was 21 days)
Population: Pharmacokinetic (PK) population included all participants who have received Tepotinib (MSC2156119J) and who had at least one blood sample drawn that provided drug concentration data for PK evaluation. Here, number analyzed signified participants evaluable at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
nanogram hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | 4440 (6.7) | 5060 (38.9)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 9
  Cycle 1 Day 15 | 15200 (18.2) | 12900 (50.4)

12. Secondary Outcome: Phase 1b: Dose Normalized Area Under the Plasma Concentration-Time Curve From Zero to Last Sampling Time at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Tepotinib
Description: Dose normalized was calculated as area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration is at or above the lower limit of quantification (LLQ) divided by the dose.
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: PK population included all participants who have received Tepotinib (MSC2156119J) and who had at least one blood sample drawn that provided drug concentration data for PK evaluation. Here, number analyzed signified participants evaluable at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
ng*h/mL/mg
  Cycle 1 Day 1 | 14.8 (6.7) | 10.1 (38.9)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 9
  Cycle 1 Day 15 | 50.7 (18.2) | 25.8 (50.4)

13. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Tepotinib
Time Frame: as for outcome 11
Population: Pharmacokinetic (PK) population included all participants who have received Tepotinib (MSC2156119J) and who had at least one blood sample drawn that provided drug concentration data for PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
nanogram hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, AUC0-inf dependent on λz was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, AUC0-inf dependent on λz was not determined.
  Cycle 1 Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, AUC0-inf dependent on λz was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, AUC0-inf dependent on λz was not determined.

14. Secondary Outcome: Phase 1b: Maximum Observed Plasma Concentration (Cmax) of Tepotinib
Description: Cmax is the maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 261 (8.4) | 278 (39.3)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 10
  Cycle 1 Day 15 | 734 (19.6) | 677 (44.6)

15. Secondary Outcome: Phase 1b: Dose Normalized Maximum Observed Plasma Concentration (Cmax) of Tepotinib
Description: Dose normalized was calculated as maximum observed plasma concentration obtained directly from the concentration versus time curve divided by dose.
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
ng/mL/mg
  Cycle 1 Day 1 | 0.871 (8.4) | 0.556 (39.3)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 10
  Cycle 1 Day 15 | 2.45 (19.6) | 1.35 (44.6)

16. Secondary Outcome: Phase 1b: Minimum Observed Plasma Concentration (Cmin) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 15 of Cycle 1 (each Cycle is 21 days)
Population: PK population included all participants who have received Tepotinib (MSC2156119J) and who had at least one blood sample drawn that provided drug concentration data for PK evaluation. Here, Overall number of participants analyzed signified participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 9
nanogram per milliliter (ng/mL) | 526 (28.0) | 435 (57.9)

17. Secondary Outcome: Phase 1b: Time to Reach Maximum Plasma Concentration (Tmax) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
hours
  Cycle 1 Day 1 | 10.0 [8.0 to 24.0] | 8.0 [8.0 to 10.0]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 10
  Cycle 1 Day 15 | 8.0 [0.48 to 8.0] | 6.1 [0.0 to 23.6]

18. Secondary Outcome: Phase 1b: Average Plasma Concentration at Steady State (Cav) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 9
nanogram per milliliter (ng/mL) | 635 (18.2) | 542 (50.7)

19. Secondary Outcome: Phase 1b: Apparent Total Body Clearance From Plasma (CL/f) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 9
Liter per hour (L/h) | 17.7 (18.2) | 34.9 (50.4)

20. Secondary Outcome: Phase 1b: Apparent Volume of Distribution During the Terminal Phase (Vz/f) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: PK population included all participants who have received Tepotinib (MSC2156119J) and who had at least one blood sample drawn that provided drug concentration data for PK evaluation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
liter
  Cycle 1 Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, VZ/F dependent on λz was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, VZ/F dependent on λz was not determined.
  Cycle 1 Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, VZ/F dependent on λz was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, VZ/F dependent on λz was not determined.

21. Secondary Outcome: Phase 1b: Apparent Volume of Distribution During the Steady State (Vss/f) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
liter
  Cycle 1 Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, VSS/F dependent on λz was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, VSS/F dependent on λz was not determined.
  Cycle 1 Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, VSS/F dependent on λz was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, VSS/F dependent on λz was not determined.

22. Secondary Outcome: Phase 1b: Apparent Terminal Elimination Rate Constant (λz) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1 per hour
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
1 per hour
  Cycle 1 Day 1 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, λz was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, λz was not determined.
  Cycle 1 Day 15 | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, λz was not determined. | NA (NA) — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, λz was not determined.

23. Secondary Outcome: Phase 1b: Apparent Terminal Half-life (t1/2) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
hours
  Cycle 1 Day 1 | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, t1/2 dependent on λz was not determined. | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, t1/2 dependent on λz was not determined.
  Cycle 1 Day 15 | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, t1/2 dependent on λz was not determined. | NA [NA to NA] — Dosing and sampling scheme in Phase Ib did not allow the reliable estimation of apparent terminal rate constant (λz), Therefore, t1/2 dependent on λz was not determined.

24. Secondary Outcome: Phase 1b: Time Prior to the First Quantifiable (Non-zero) Concentration (Tlag) of Tepotinib
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 Cycle 1 (each Cycle is 21 days)
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 12
hours | 0.53 [0.52 to 0.55] | 0.50 [0.25 to 1.0]

25. Secondary Outcome: Phase 1b: Percentage Peak-Trough Fluctuation (PTF) Post First Dose of Tepotinib
Description: The peak trough fluctuation within complete dosing interval at steady state, calculated as PTF (%) = ([Cmax - Cmin]/Cav ) multiplied by 100
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage fluctuation
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 9
percentage fluctuation | 31.5 (30.5) | 35.9 (44.1)

26. Secondary Outcome: Phase 1b: Accumulation Ratio of Cmax (Racc (Cmax))
Description: Accumulation ratio for Cmax was calculated as Cmax, after dosing on Day 15 divided by Cmax, after dosing on day 1 of cycle 1.
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 10
ratio | 2.81 (24.1) | 2.32 (23.0)

27. Secondary Outcome: Phase 1b: Accumulation Ratio of AUC (Racc (AUC)
Description: Accumulation ratio for AUC was calculated as AUC, after dosing on Day 15 divided by AUC, after dosing on day 1 of cycle 1.
Time Frame: Pre-dose and at 0.25, 0.5, 1, 2, 4, 8, 10, and 24 hours post-dose; Day 1 and Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 16
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg
Number analyzed (Participants) | 3 | 9
ratio | 3.43 (22.6) | 2.51 (22.0)

ADVERSE EVENTS:
Time Frame: From date of randomization up to 1369 days
Arm/Group | Phase 1b: Tepotinib 300 mg | Phase 1b: Tepotinib 500 mg | Phase 2: Tepotinib 500 mg
All-Cause Mortality (participants affected / at risk) | 3/4 | 11/13 | 40/49
Serious Adverse Events (participants affected / at risk) | 2/4 | 5/13 | 21/49
Other Adverse Events (participants affected / at risk) | 4/4 | 12/13 | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Tepotinib 300 mg (N=4) | Phase 1b: Tepotinib 500 mg (N=13) | Phase 2: Tepotinib 500 mg (N=49)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Disease progression (General disorders) | 1 | 1 | 7
Localised oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 2 | 1
Discomfort (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Tepotinib 300 mg (N=4) | Phase 1b: Tepotinib 500 mg (N=13) | Phase 2: Tepotinib 500 mg (N=49)
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 7
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 4
Ascites (Gastrointestinal disorders) | 0 | 2 | 15
Constipation (Gastrointestinal disorders) | 2 | 0 | 9
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 16
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Gastric varices (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 11
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 7
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 2 | 15
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 10
Generalised oedema (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 1 | 2
Oedema (General disorders) | 0 | 0 | 3
Oedema peripheral (General disorders) | 3 | 10 | 32
Pyrexia (General disorders) | 1 | 1 | 4
Pain (General disorders) | 0 | 1 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 2
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 4
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 2
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0
Angular cheilitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 4 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 6
Blood alkaline phosphatase increased (Investigations) | 2 | 2 | 5
Blood bilirubin increased (Investigations) | 0 | 1 | 5
Blood creatinine increased (Investigations) | 1 | 2 | 7
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 2 | 3
International normalised ratio increased (Investigations) | 0 | 0 | 2
Lipase increased (Investigations) | 1 | 1 | 5
Prothrombin time prolonged (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Urobilinogen urine increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 1
Amylase increased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 8
Cell death (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 5
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 2
Depressed mood (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 3
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 2 | 0
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1
Ketonuria (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT02115373/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT02115373/SAP_001.pdf